CLINICAL TRIAL: NCT05658016
Title: A Phase 2a, Multi-center, Placebo-Controlled, Randomized, Assessor-blind Study to Assess the Safety & Efficacy of Parenteral TK-90 or Parenteral TK-90 Placebo to Patients Receiving Radiotherapy for Non-Metastatic Squamous Cell Carcinoma of Head and Neck.
Brief Title: Phase 2a Study to Evaluate Suppression of Radiotherapy-induced Mucositis by TK112690
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tosk, Inc. (Industry)
Collaborators: SIRO Clinpharm Private Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CLP-2690-0004
Record Dates: First submitted 2022-12-01; First posted 2022-12-20 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Mucositis
Keywords: Mucositis; Uridine Phosphorylase Inhibitor; Head and Neck Cancer; Radiation
MeSH Terms: conditions — Mucositis; Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: A total of 24 patients will be enrolled into one of 2 different: TK112690 treated or placebo treated.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study will be partially blinded. The patient and investigator as well as site personnel will be blinded as to whether TK-90 or TK-90 placebo is administered. The CRO, sponsor, and site pharmacist will know whether the patient was administered active drug or TK-90 placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TK112690 (Experimental): TK112690 treatment
  Interventions: Drug: TK-112690
- Placebo (Placebo Comparator): TK112690 formulation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TK-112690 — TK112690 treatment Pre & Post Radiation
  Arms: TK112690
Drug: Placebo — TK112690 Placebo treatment Pre & Post Radiation
  Arms: Placebo

SUMMARY:
Patients expected to receive a continuous course of radiation as single daily fractions of 2.0 Gy treatment with a cumulative radiation dose of 70 Gy. The radiation can be 2DRT, 3DRT,IMRT etc. Prior to each radiation treatment the patients will receive a one-hour infusion of TK-90 or equivalent TK-90 placebo depending on randomization. 6 Hours after the completion of TK-90 infusion or TK-90 placebo dose, the patients will receive another identical TK-90 or TK-90 placebo treatment depending on randomization. This treatment cycle will continue for 7 weeks. The TK112690 dose will be 45 mg/kg.

DETAILED DESCRIPTION:
Patients expected to receive a continuous course of radiation as single daily fractions of 2.0 Gy treatment with a cumulative radiation dose of 70 Gy. The radiation can be 2DRT, 3DRT,IMRT etc. Prior to each radiation treatment the patients will receive a one-hour infusion of TK-90 or equivalent TK-90 placebo depending on randomization. 6 Hours after the completion of TK-90 infusion or TK-90 placebo dose, the patients will receive another identical TK-90 or TK-90 placebo treatment depending on randomization. This treatment cycle will continue for 7 weeks. The TK112690 dose will be 45 mg/kg.

* 24 patients will be randomized equally into 2 different groups: TK-90 treated or TK-90 placebo treated.
* Screening must be completed within 2 weeks.
* The treatment period for the study is 7 weeks.
* Study follow-up will be scheduled post two weeks of completion of last dose of radiation or early termination through up to 4 weeks.
* Blinding: The study will be partially blinded. The patient and investigator as well as site personnel will be blinded as to whether TK-90 or TK-90 placebo is administered. The CRO, sponsor, and site pharmacist will know whether the patient was administered active drug or TK-90 placebo.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet ALL of the following criteria at the time of screening unless otherwise specified:

  1. Patient must sign study specific informed consent prior to study entry.
  2. Male or Female patient aged 18 - 75 years.
  3. Pathologically (histologically or cytologically) proven (from primary lesion and/or lymph nodes) diagnosis of squamous cell carcinoma of the oral cavity (Refer Definition in 10.13.1), oropharynx or hypopharynx.
  4. Patients must have at least 1 mucosal site of the oral cavity/oropharynx/hypopharynx mucosa assessable by visual transoral inspection that will receive cumulative radiation dose of 70 Gy.

     Note: Unavoidable doses of at least 60 Gy, to include entrance, exit, and scatter doses, still constitutes planned radiation.
  5. Patients with tumors of the larynx or hypopharynx are eligible only if it is anticipated that at least 1 index site in the oral cavity/oropharynx/hypopharynx mucosa (Refer section 10.13.1) will receive cumulative radiation dose of 70 Gy.
  6. Selected Stage I to III or IVA-B per AJCC, Cancer Imaging Manual, 8th edition, at study entry, including no distant metastases other than non- metastatic SCCHN, based upon the following minimum diagnostic workup:

     * History/physical examination, including documentation of tobacco/alcohol use and current medications (including opioids/dosing), within 8 weeks prior to randomization.
     * Chest CT scan within 8 weeks prior to randomization.
     * MRI or CT scan with contrast of tumor site within 8 weeks prior to randomization.
  7. Mucositis Grade ≤ 1 per WHO Scale and Xerostomia of Grade ≤ 2 per CTCAE version 5.0
  8. ECOG Performance Status ≤ 2.
  9. Adequate bone marrow function as per CTCAE V 5, defined as follows (within 2 weeks prior to randomization):

     * Absolute neutrophil count ≥ 1500cells/mm3 based upon CBC/differential obtained within 2 weeks prior to randomization.
     * Platelets ≥ 100,000 cells/mm3 based upon CBC/differential obtained within 2 weeks prior to randomization.
     * Hemoglobin ≥ 8.0 g/dl based upon CBC/differential obtained within 2 weeks prior to randomization (Note: The use of transfusion or other intervention to achieve Hgb> 8.0 g/dl is acceptable).
  10. Adequate hepatic function with bilirubin ≤ 1.5 x upper-normal limit (ULN), AST or ALT ≤3 x ULN within 2 weeks prior to randomization.
  11. Adequate renal function with serum creatinine < 1.5 mg/dl and creatinine clearance (CrC) ≥ 50 ml/min determined by 24-hour collection or estimated by Cockcroft-Gault formula. CrC male = [(140 - age) x (wt in kg)] / [(Serum Cr mg/dl) x (72)]. CrC female = 0.85 x (CrCl male) within 2 weeks prior to randomization.
  12. Normal serum calcium or normal corrected serum calcium within 2 weeks prior to randomization; formula for corrected calcium if albumin valued is below normal range: Corrected calcium (mg/dl) = (4 - [Patient's albumin (g/dl)] x 0.8) + Patient's measured calcium (mg/dl).
  13. Negative serum pregnancy test for women of childbearing potential.
  14. Women of childbearing potential and male participants with female partners of childbearing potential must practice adequate contraception.

Exclusion Criteria:

Patients who meet any of the following criteria at the time of screening will be excluded:

1. Stage IVC (Any T, Any N, M1) per AJCC Cancer Staging Manual. 8th ed, or distant metastases at protocol study entry other than metastatic SCCHN.
2. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years.
3. Patients who have not fully recovered after prior surgery. (Patients who have had prior surgery and have fully recovered and patients who may have surgery in the future are eligible.).
4. Severe, active co-morbidity, defined as follows:

   * Symptomatic and/or uncontrolled cardiac disease, New York Heart Association Classification III or IV.
   * Transmural myocardial infarction within the last 6 months.
   * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of screening.
   * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of screening.
   * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects.
   * Patients known to be sero-positive for human immunodeficiency virus (HIV), hepatitis B (HBV), hepatitis C (HCV).
5. Collagen vascular disease, such as scleroderma.
6. Previous treatment with palifermin or other keratinocyte growth factors, such as velafermin or repifermin, within 28 days of randomization.
7. Any prohibited therapy 2 weeks prior to randomization (see Section 8.4).
8. Pregnancy, breast feeding or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception.
9. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
10. Known hypersensitivity study medication or excipients in the formulation.
11. Any illness or medical conditions that are unstable or could jeopardize the safety of the patient and his/her compliance in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Mucositis | 7 weeks
  * SOM (Severe Oral Mucositis) - Comparison of incidences of Grade 3 or 4 mucositis (WHO scale) in the treatment and placebo groups.
  * Duration of SOM (Severe Oral Mucositis). Days patients suffer Grades 3 and 4 oral mucositis measured by WHO scale from the start of treatment.
  * Calculate Number of days from the first occurrence of WHO Grade 3 or 4 oral mucositis through the first occurrence of non-severe (≤ Grade 2) without a subsequent instance of ≥ Grade 3 oral mucositis.
  * Subjects with complete study follow-up for SOM who do not develop severe oral mucositis (grade 0-2) will be considered to have duration of 0 days.

SECONDARY OUTCOMES:
Secondary efficacy/outcome mucositis | 7 weeks
  * Mucositis status in the patients will also be evaluated using two different published and validated mucositis scales: NCI/CTCAE/mucositis, and PROMS.
  * Comparison of WHO scale values of treated patients at each point of evaluation.
  NCI/CTCAE=National Cancer Institute/Common Terminology Criteria for Adverse Events and WHO=World Health Organization PROMS=Patient Reported oral Mucositis Symptom Scale
  As per WHO:Grade 0 to Grade 5 & NCI CTCAE: Grade 1 to Grade 5
Incidence Adverse Events That Are Related to Treatment | 7 Weeks
  Tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Emile Youssef, MD, PhD, Study Director — Tosk, Inc.
Locations (5):
- India (5):
  - Sher-I-Kashmir Institute of Medical Sciences, Srinagar, Jammu and Kashmir
  - Bangalore Medical college and Research Institute, Bangalore, Karnataka
  - Saveetha Medical College and Hospita, Chennai, Tamil Nadu
  - Apex Hospital, Varanasi, Uttar Pradesh
  - Netaji Subhash Chandra Bose Hospital, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: No